CLINICAL TRIAL: NCT05837715
Title: Investigation of the Effects of Cervical Stabilization Exercises and Vibration Application to the Cervical Region on Motor Symptoms and Sensory Profile in Individuals With Parkinson's Disease
Brief Title: Effects of Cervical Stabilization Exercises and Vibration Application in Individuals With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Emine Nur Demircan, Physiotherapist (PhD student in Hacettepe University), Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: stabilization and vibration
Record Dates: First submitted 2023-04-05; First posted 2023-05-01 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Parkinson Disease
Keywords: cervical; stabilization exercises; vibration; motor symptoms; impaired sensation; Parkinson disease
MeSH Terms: conditions — Parkinson Disease; Hypesthesia | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- stabilization group (Experimental): cervical stabilization exercises
  Interventions: Device: Chattanooga Stabilizer pressure biofeedback
- vibration group (Experimental): vibration application to the cervical region
  Interventions: Device: VibraSens - Focal Vibration Therapy (TechnoConcept - France)
- telerehabilitation group (Experimental): online exercise method
  Interventions: Other: Telerehabilitation

INTERVENTIONS:
Device: Chattanooga Stabilizer pressure biofeedback — Stabilization exercises, which form the basis of spinal stabilization training, increase the strength and endurance of the postural and stabilizer muscles by using the basic principles of motor learning, and improve balance control in stable and unstable positions.
  In addition, stabilization exercises include kinesthetic training and functional training.
  Spinal stabilization training is very important for proper control of extremity movements.
  It is also an important factor in the formation of proper spinal posture and the neutral position required for the spine.
  In cervical region problems, cervical stabilization exercises that activate the deep neck flexors (longus colli and longus capitis) can be applied.
  Cervical stabilization training improves the cervical proprioception sense as well as strength and endurance, thereby reducing joint position sense error.
  Arms: stabilization group
Device: VibraSens - Focal Vibration Therapy (TechnoConcept - France) — Vibration applications have also started to be used for treatment purposes. Therapeutic vibration produces minor changes in skeletal muscle length. Vibrations elicit a response called the "tonic vibration reflex", which includes activation of muscle spindles, neural signals by Ia afferents, and activation of muscle fibers via large α-motor neurons. The tonic vibration reflex can also cause an increase in activation of motor units through activation of muscle spindles and polysynaptic pathways. It is well known that the input of the proprioceptive pathways (Ia, IIa and possibly IIb) plays an important role in the production of isometric contractions. The increase in isometric strength after application of vibration with extensive sensory stimulation may be the result of more efficient use of the positive proprioceptive feedback loop. It can be predicted that the increased muscle strength after vibration application is due to neural adaptation.
  Arms: vibration group
Other: Telerehabilitation — Telerehabilitation is a method that aims to provide rehabilitation to patients/clinicians by reducing obstacles such as distance, time and cost by using information and communication technologies. Telerehabilitation enables patients who cannot access rehabilitation due to geographic, economic or physical disabilities to benefit from rehabilitation services. The COVID-19 pandemic has highlighted the importance of telerehabilitation practices. In order to minimize the risk of transmission in the COVID-19 pandemic, the physical activity levels of individuals have decreased and their access to rehabilitation services has been restricted by the restriction of social life.
  Arms: telerehabilitation group

SUMMARY:
Parkinson's disease (PD) is the second most common neurodegenerative disease that causes a progressive decrease in motor functions, which is caused by the influence of dopaminergic pathways in the substantia nigra (SN). Motor and non-motor symptoms seen in PD seriously affect patients negatively.

Proprioception, which is one of the deep senses, is known to help maintain body verticalization in the sense of posture and movement and has a primary importance in the regulation of motor activities. Depending on the progression of the disease, flexion of the body is triggered as a result of the deterioration of proprioception over time. It is suggested that the losses in proprioception may result from the inability to properly regulate motor control and body reflexes. Therefore, the assessment of proprioception plays an important role in assessing changes in postural instability, gait and fall risk.

It is said that while peripheral muscle feedback is preserved in Parkinson's patients, there is deterioration in integration in the central. Changes in the supraspinal processing of proprioceptive input in PD have been demonstrated by analyzing the effect of mechanical vibration applied to the tendon of a stretched muscle during voluntary movements. Vibrator stimulation activates muscle spindle afferents, particularly primary endings. It is also stated that muscle feedback is not only related to the movement performed, but also to the response induced by vibration.

In line with this information, vibration applications have been added to the treatment of PD in recent years with the aim of stimulating postural adjustments through the application of an external proprioceptive input.

It is selectively used in neurological rehabilitation because of the effect of local vibration training on spinal excitability. When the literature is examined, it has been determined that the studies on the effects of local vibration applied to the neck region on posture, balance, proprioception and other sensory profiles are insufficient, especially in individuals with Parkinson's disease.

In this project, it is aimed to guide professionals working with Parkinson's disease in the management of this disease by determining the effects of cervical stabilization and local vibration application to the cervical region on motor symptoms and sensory profile in individuals with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Being diagnosed with idiopathic Parkinson's Disease
2. To be between the ages of 40-80,
3. The duration of the disease is 3 years or more,
4. Being between stage 2 and 3 according to the Modified Hoehn-Yahr Staging Scale [Modified Hoehn & Yahr Staging Scale: This scale examines the disease in 5 stages (82). These phases are:

   * Stage 1: Unilateral tremor, rigidity, akinesia or postural instability.
   * Stage 1.5: Unilateral and axial involvement.
   * Stage 2: Postural abnormalities with or without axial signs such as bilateral tremor, rigidity, akinesia or bradymia, swallowing difficulties, axial rigidity (especially neck), forward-bending posture, slow or shuffling gait, and general stiffness
   * Stage 2.5: Mild bilateral disease with improvement in tensile test
   * Stage 3: In addition to the findings in Stage 2, the patient has balance disorder, but the patient can perform all activities independently.
   * Stage 4: The patient needs help in some or all activities of daily living.
   * Stage 5: The patient is wheelchair or bed-bound].
5. A score of 24 or higher on the Standardized Mini-Mental test, Standardized Mini-Mental Test: There are 19 items in this test, which consists of 5 main sections: orientation, recording memory, attention and calculation, recall and language. The total score of the test is evaluated out of 30 and 24 points are accepted as the threshold value for the diagnosis of mild dementia (83).
6. Not have any additional orthopedic, vestibular and/or neurological disease other than Parkinson's Disease that will affect muscle strength, sense, balance and coordination.
7. Not having undergone any surgical procedure that may affect the stabilization of the musculoskeletal system of the spinal column and lower extremity.

Exclusion Criteria:

1. Having a pacemaker,
2. Having a psychiatric disease, uncontrollable dyskinesia or motor fluctuations, postural hypotension that may affect balance, vision problems,
3. Individuals with orthopedic problems that may cause limitation of movement and inflammatory arthritis (such as fractures, osteoporosis, osteomyelitis) will be excluded from the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-30 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
Change of Recording Demographic Data | baseline - change at 6 weeks - 4 weeks later
  At the beginning of the study, demographic characteristics of all participants such as age, gender, dominant hand and dominant foot, CV and family history will be recorded. In addition, disease-related information such as the time of diagnosis, the dominant side, the side of the disease, and the drugs used will also be recorded.
Change of Movement Disorders Association, Unified Parkinson's Disease Rating Scale | baseline - change at 6 weeks - 4 weeks later
  The scale consists of 4 subheadings, the 1st part being non-motor problems, the 2nd part motor problems, the 3rd part motor examination and the 4th part motor complications. In the scale consisting of 50 items, each question has five answer options between 0 and 4 points.
Change of cervical region joint position sense | baseline - change at 6 weeks - 4 weeks later
  The subject sits upright in a comfortable position with arms at the side. First of all, the active maximum range of motion of the subjects in 6 different positions is determined separately, and 65 percent of this value is calculated. The subject is then asked to close his eyes and the subject's head is slowly and passively brought to the point previously determined by the physiotherapist. The head of the subject is held for three seconds at the passively brought point and asked to feel the joint position. Then, the subject's head is brought back to the neutral position and asked to actively bring it to that point, which is passively brought. The difference between the point where the phenomenon comes from and the previously determined reference point is calculated and determined as the insertion position sense error.
Change of Vibration Sense | baseline - change at 6 weeks - 4 weeks later
  Vibration sense will be evaluated using tuning fork with a frequency of 128-Hz. After explaining how the test will be done and what is requested from the patient, the tuning fork to be used during the test will be placed on the patient's areas to be tested in order for the patient to feel and learn the vibration.
Change of Light touch-Pressure Sense | baseline - change at 6 weeks - 4 weeks later
  With the Semmes Weinstein Monofilament Test, it will be applied to the tips of the thumbs in the hand and under the soles of the feet.) and the Sense of Steregnosis will be evaluated.
Change of Craniocervical Flexion Strength | baseline - change at 6 weeks - 4 weeks later
  This test tests the activation and endurance of the deep neck flexors. It is performed with the individual lying in the supine hook position and the neck in a neutral position. The uninflated pressure sensor is placed between the projection of the earlobe and the chin and inflated to 20 mmHg. The person is asked to do the movement lightly and slowly (as if to nod, as if to say yes) and look towards their eyes and feet. Activation score is calculated based on the pressure level that the person is able to achieve and can do 10 repetitions for a 10-second period and deep cervical flexor recorded as a measurement of the strength of the muscles.
Change of Endurance Cervical Flexor Muscles | baseline - change at 6 weeks - 4 weeks later
  The case is performed in the supine hooked position, with the hands free on the abdomen. The subject is asked to raise his head slightly at a height of about 2 cm, and after this position is taught, he is asked to do a slight (30%) craniocervical flexion as if he were saying yes. The time it takes to maintain the position while maintaining the craniocervical flexion movement is recorded in seconds.
Change of Respiratory Muscle Strength | baseline - change at 6 weeks - 4 weeks later
  It will be evaluated with the "Respiratory pressure meter - RP Check" device.
Change of Balance | baseline - change at 6 weeks - 4 weeks later
  It will be evaluated with the TecnoBody device.
Change of Functional Reach Test | baseline - change at 6 weeks - 4 weeks later
  Test is a dynamic test used to evaluate postural control. Values less than 25.4 cm indicate increased risk of falling (92), and values less than 15.24 cm indicate physical frailty.
Change of New York Posture Analysis | baseline - change at 6 weeks - 4 weeks later
  In this evaluation system, postural changes in 13 different parts of the body are examined. Accordingly, five points are given if the person's posture is correct, three points if moderately impaired, and one point if severely impaired. The total score obtained as a result of the test is a maximum of 65 and a minimum of 13.
Change of Basic Digital Inclinometer - Inclinometer | baseline - change at 6 weeks - 4 weeks later
  An "inclinometer" device will be used in the evaluation of thoracic kyphosis and lumbar lordosis. In order to determine the thoracic kyphosis, the "inclinometer" will measure the spinous processes of the C7-T1 and T12-L1 vertebrae, and the degrees found will be summed and the degree of kyphosis will be calculated. In order to determine the lumbar lordosis, measurements will be made between the spinous processes of the T12-L1 and S2-S3 vertebrae and the degree of lordosis will be calculated by adding the degrees found.
Change of Baseline Inclinometer | baseline - change at 6 weeks - 4 weeks later
  A "Baseline Scoliometer" device will be used to evaluate the cervical curvature of the cases. For cervical lordosis, the graduated dial will be set parallel to the ground. The top bar of the device will be locked and inserted into the spinous process of the C4 vertebra. The lower bar will be adjusted in height so that it is in the spinous process of the C7 vertebra. The lower bar will be loosened until the indicator shows zero degrees, locked at the point where it points zero, and the measurement will be recorded in cm.
Change of Freezing Scale While Walking | baseline - change at 6 weeks - 4 weeks later
  On a 6-item scale, it is questioned whether frostbite occurs during activities such as walking and turning, and in case of frostbite, the severity, frequency and duration of frostbite are recorded. Items 1, 2, 4, 5 and 6 of the scale are related to the experiences of the patients, especially in the last week; The third item defines the frequency of frostbite seen in patients.

SECONDARY OUTCOMES:
Change of Timed Get Up and Go Test | baseline - change at 6 weeks - 4 weeks later
  In this test, which is conducted to evaluate dynamic balance and functional mobility, the individual will be asked to get up from a chair with back support and without arm support, walk a three-meter distance, turn around, and sit back in the chair. The elapsed time will be recorded in seconds. Three repetitions will be performed and the best result will be recorded. The number of steps taken will also be recorded as cadence.
Change of 2 Minute Walk Test | baseline - change at 6 weeks - 4 weeks later
  The 2-Minute Walk Test (2MWT) is a valid and reliable measure of mobility that assesses walking endurance for individuals with PD. The 2MWT can detect that people with PD walk less than controls of the same age. For this study, subjects will be instructed to walk on a flat surface and "cover as much distance as possible" for 2 minutes.
Change of Parkinson's Disease Questionnaire-39 | baseline - change at 6 weeks - 4 weeks later
  This scale, which evaluates the daily living activities of Parkinson's patients, consists of mobility, daily living activity, emotional well-being, stigma, social support, cognition, communication, and physical discomfort. The total score obtained from the scale ranges from 0 to 100. As the score increases, the quality of life worsens.

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet